CLINICAL TRIAL: NCT02864199
Title: Non-Randomized, Multicenter Study to Evaluate the Pharmacokinetics and Safety of Peginterferon Alfa-2a and Copegus Combination Therapy After Single and Multiple Doses in Patients With Chronic Hepatitis C and Moderate Renal Impairment, Severe Renal Impairment, or End-Stage Renal Disease Undergoing Hemodialysis
Brief Title: A Study of Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) Combination Therapy in Participants With Chronic Hepatitis C (CHC) and Various Degrees of Renal Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP17355
Record Dates: First submitted 2016-08-09; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (4):
- Group A: Moderate Renal Impairment (Experimental): Participants with CrCl 30 to 50 mL/min will receive 12 weeks of peginterferon alfa-2a, 180 micrograms (mcg) via subcutaneous (SC) injection once weekly, in combination with ribavirin, 600 milligrams (mg) orally (PO) daily in two divided doses. Those with Genotype 2 or 3 disease may receive an additional 12 weeks of the same regimen, and those with another genotype may receive an additional 36 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group B: Severe Renal Impairment (Experimental): Participants with CrCl <30 mL/min will receive 12 weeks of peginterferon alfa-2a, 180 mcg via SC injection once weekly, in combination with ribavirin, 400 mg PO daily in two divided doses. Those with Genotype 2 or 3 disease may receive an additional 12 weeks of the same regimen, and those with another genotype may receive an additional 36 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group C: Hemodialysis/ESRD (Experimental): Participants requiring hemodialysis will receive 12 weeks of peginterferon alfa-2a, 135 mcg via SC injection once weekly, in combination with ribavirin, 200 mg PO every morning. Those with Genotype 2 or 3 disease may receive an additional 12 weeks of the same regimen, and those with another genotype may receive an additional 36 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group D: Normal Renal Function (Experimental): Participants with CrCl >80 mL/min will receive 12 weeks of peginterferon alfa-2a, 180 mcg via SC injection once weekly, in combination with ribavirin, 800 to 1200 mg PO daily in two divided doses. Those with Genotype 2 or 3 disease may receive an additional 12 weeks of the same regimen, and those with another genotype may receive an additional 36 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a will be administered for 12 to 48 weeks. The dose will range from 135 mcg (Group C) to 180 mcg (Groups A, B, and D) once weekly via SC route.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin will be administered for 12 to 48 weeks. The total daily dosage will range from 200 mg (Group C) to 1200 mg (Group D), depending upon CrCl and participant-specific factors.
  Other Names: Copegus

SUMMARY:
This study will evaluate the pharmacokinetics (area under the curve [AUC], maximum concentration [Cmax], and other parameters) and tolerability of peginterferon alfa-2a and ribavirin combination therapy following single and multiple doses in participants with CHC infection and moderate to severe renal impairment or end-stage renal disease (ESRD) receiving hemodialysis. The anticipated time on study treatment is up to 48 weeks, and the target sample size is 48 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years of age
* CHC infection as shown on enzyme-linked immunosorbent assay (ELISA) and radioimmunoblot assay (RIBA) or quantifiable hepatitis C virus (HCV) ribonucleic acid (RNA) greater than (>) 2000 copies per milliliter (copies/mL)
* Use of two forms of contraception during study and 6 months after the study in both men and women
* Normal renal function (creatinine clearance [CrCl] >80 milliliters per minute [mL/min]), moderate renal impairment (CrCl 30 to 50 mL/min), severe renal impairment (CrCl less than [<] 30 mL/min), or ESRD requiring hemodialysis
* Patients with ESRD must have been undergoing hemodialysis for at least 2 months

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Male partners of women who are pregnant
* Conditions associated with decompensated and/or chronic liver disease
* Human immunodeficiency virus (HIV) infection
* Interferon or ribavirin treatment within the previous 3 months
* Poor hematologic function, including unstable hemoglobin
* Significant comorbidity or severe illness which would make the participant unsuitable for the study
* Acute renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cmax of peginterferon alfa-2a | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
CL/F of ribavirin | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
Percentage of participants with undetectable HCV RNA level | Week 12
Cmax of ribavirin | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
AUC of ribavirin | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
AUC of peginterferon alfa-2a | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
Clearance (CL/F) of peginterferon alfa-2a | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12

SECONDARY OUTCOMES:
Time of maximum concentration (Tmax) of peginterferon alfa-2a | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
Tmax of ribavirin | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
Plasma concentration of ribavirin | Pre-dose (0 hours) and 0.5, 1, 3, 5, 8, 12, 24, 72, 120, and 168 hours post-dose during Weeks 1 and 12
Percentage of participants with adverse events (AEs) | From Baseline to Week 12 (or up to Week 48 if treatment continued)
Percentage of participants with a dose modification or premature withdrawal for safety reasons | From Baseline to Week 12 (or up to Week 48 if treatment continued)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (17):
- United States (12):
  - Birmingham, Alabama
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Kansas City, Missouri
  - St Louis, Missouri
  - New York, New York
  - Syracuse, New York
  - Cleveland, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Galveston, Texas
- São Paulo, Brazil
- Marseille, France
- New Zealand (2):
  - Christchurch
  - Riccarton, Christchurch
- Huddinge, Sweden